CLINICAL TRIAL: NCT06402903
Title: Physiotherapy in Patients in a Cardiac Intensive Care Unit. A Retrospective Cohort Study
Brief Title: Physiotherapy in Patients in a Cardiac Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Ruben Cuesta Barriuso, Principal Investigator, University of Oviedo
Other Study IDs: FisCard
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Surgery Patients
Keywords: Physiotherapy; Intensive Care Unit; Postoperative complications prevention; Cardiac surgery
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observacional group: The data will be collected in April 2024 at the Physical Medicine and Rehabilitation Service of the Central University Hospital of Asturias (HUCA), belonging to Health Area IV of the Health Service of the Principality of Asturias.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — The clinical, post-surgical and anthropometric variables of the patients, as well as the time spent in the Intensive Care Unit and on the hospital ward (in days) were collected in the Clinical Histories.
  The collection of data from the Clinical Histories will be carried out by the principal investigator, an employee of the Hospital Universitario Central de Asturias, in accordance with current data protection regulations, scrupulously complying with the anonymous collection of clinical data, and without collecting any data that could allow the identification of the patients whose data were collected.
  The data from the Clinical Histories will be exported to an Excel file which will subsequently be anonymised. Access to the Excel file will require a password access that will be managed from a computer of the University of Oviedo (Department of Surgery and Medical-Surgical Specialties).

SUMMARY:
Background. Cardiovascular diseases are a major cause of morbidity and mortality. The management of these patients requires multidisciplinary therapeutic approaches. Physiotherapy plays a fundamental role in the postoperative management of patients undergoing cardiac surgery.

Objective: To analyse the relationship between the administration of a physiotherapy intervention and the time spent in the cardiac ICU and on the ward.

Method. Retrospective cohort study. The medical records of 110 patients undergoing cardiac surgery who received a Physiotherapy intervention during their stay in the Intensive Care Unit will be analysed. Data will be collected from patients admitted to the cardiac ICU in 2023. The variables assessed will be: length of stay in ICU and hospital admission (days), age (years completed), weight (kg) and sex. A one-factor analysis of variance will be performed to calculate the association between the variables and a linear regression analysis will be used to describe the hospital stay variables as a function of the other predictor variables.

Expected outcomes. Physiotherapy treatment in an Intensive Care Unit improves ICU and hospital stay times in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cardiac pathology
* Undergoing cardiac surgery at the Hospital Universitario Central de Asturias between 1 January and 31 March 2023
* In the postoperative phase in the Intensive Care Unit and subsequently on transfer to the ward, they received physiotherapy treatment or not.
* That the period of stay in the ICU was less than 30 days.

Exclusion Criteria:

* Patients with comorbidities prior to surgery that hindered independence from third parties in the performance of activities of daily living and ambulation; iii) patients with previous cardiac surgeries; and iv) patients whose study variables were not fully recorded in the Medical History.
* Patients with previous cardiac surgeries
* Patients whose study variables were not fully recorded in the Clinical History.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The data will be collected in May 2024 at the Physical Medicine and Rehabilitation Service of the Hospital Universitario Central de Asturias (HUCA), belonging to the Health Area IV of the Health Service of the Principality of Asturias.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Assess length of stay in the Intensive Care Unit | Screening visit
  This period shall be calculated (in days) by subtracting the date of admission to the Intensive Care Unit from the date of discharge from the Intensive Care Unit.
Assess time from hospital admission to medical discharge | Screening visit
  This period shall be calculated (in days) by subtracting the date of admission to the Intensive Care Unit from the date of discharge.

SECONDARY OUTCOMES:
Assess the age | Screening visit
  This quantitative variable will indicate the age of the patients (in years of age) at the time of admission to the Intensive Care Unit.
Assess the gender | Screening visit
  This dichotomous variable (Female / Male) will indicate the sex of the patient at the time of admission to the Intensive Care Unit.
Assess the weight | Screening visit
  The weight at the time of the patient's admission to the hospital will be assessed (in kg)
Assess the administration of a physiotherapy intervention | Screening visit
  This dichotomous variable (Yes / No) will indicate whether the patient has received physiotherapy intervention during his/her stay in the Intensive Care Unit.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain